CLINICAL TRIAL: NCT06123325
Title: Impact of Observation Versus Treatment on The Psychiatric and Mental Outcomes of Patients With Unruptured Intracranial Aneurysms
Brief Title: Psychiatric Outcomes of Unruptured Intracranial Aneurysms (POUIA)
Acronym: POUIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: The Bee Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-15285
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Anxiety Depression; Aneurysm Cerebral; Mental Health Wellness 1
Keywords: Cerebral aneurysm; Anxiety; Depression; Endovascular; Clipping
MeSH Terms: conditions — Intracranial Aneurysm; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Controlled, non-randomized, prospective cohort study with parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Patients with unruptured intracranial aneurysms, opting for active intervention undergo microsurgical clipping or endovascular therapy to preemptively secure the aneurysm and prevent rupture.
  Interventions: Procedure: Clipping; Procedure: Endovascular embolization
- Observation group (Other): Patients with unruptured intracranial aneurysms, opting for conservative management undergo regular monitoring with serial imaging to track aneurysm stability, deferring interventional treatment unless changes indicate an increased risk of rupture.
  Interventions: Diagnostic Test: Surveillance imaging

INTERVENTIONS:
Procedure: Clipping — Microsurgical clipping of intracranial aneurysms involves craniotomy to access the brain, locating the aneurysm, and placing a small metal clip across its neck, thereby isolating it from normal blood circulation to prevent rupture.
  Arms: Treatment group
Procedure: Endovascular embolization — Any endovascular embolization of intracranial aneurysms that involves navigating microcatheters through the vascular system to the site of the aneurysm and deploying materials like coils, flow-diverting stents, or endosaccular flow disruptors to occlude the aneurysm and reduce the risk of rupture.
  Arms: Treatment group
Diagnostic Test: Surveillance imaging — Surveillance imaging for brain aneurysms is a diagnostic approach that uses imaging techniques such as MRI, MRA, CTA, or DSA to regularly monitor the status of detected brain aneurysms. The goal is to track changes in the aneurysm's size, shape, or structure over time, which may indicate an increased risk of rupture. This ongoing assessment helps healthcare providers decide whether to continue monitoring or to consider treatment options, such as surgical clipping or endovascular coiling, based on the aneurysm's characteristics and the patient's risk factors.
  Arms: Observation group

SUMMARY:
The impact of cerebrovascular procedures on patients experiencing anxiety and depression is not well studied despite the high prevalence of these mental health disorders. Unruptured Intracranial aneurysms (UIAs) have a prevalence of approximately 3% and an annual risk of 1-2% in the general population. Despite the high risk of fatality following aneurysm rupture with a rate of 40-50%, the overall aneurysm growth and rupture risks are rare (less than 3% per aneurysm per year) and many patients can be observed with serial follow-up imaging over years. Nevertheless, due to the gravity of the bad consequences of aneurysm rupture, simply informing many patients of UIA diagnosis has been found to result in worse outcomes of health-related quality of life. This study aims to investigate the impact of awareness of untreated UIA on the patients' mental health utilizing the Hospital Anxiety and Depression Scale (HADS) tool.

DETAILED DESCRIPTION:
This is a controlled, non-randomized, prospective cohort study with parallel arms of treatment arm with microsurgical and endovascular treatment and comparison control arm with conservative management/observation of UIA. The goal of this study is to investigate the impact of the awareness of an untreated UIA on the psychiatric and mental status of the patients enrolled in the control arm compared to patients with a treated UIA. All patients presenting to the outpatient clinic upon the initiation of the trial and for 2 years ahead with UIA diagnosed on any of the angiographic imaging modalities including Computed Tomography Angiography (CTA), Magnetic Resonance Angiography (MRA), and Digital Subtraction Angiogram (DSA) will be included.

ELIGIBILITY:
Inclusion Criteria:

* Unruptured intracranial aneurysms (UIA)
* mRS scores between 0-1
* Observation Group: All patients with UIAs that are eligible for conservative management

  1. Specific locations that are not good candidates for interventional treatment, such as cavernous internal carotid artery and very distally located aneurysms
  2. Aneurysm size (largest dimension) is less than 4 mm
* Treatment Group: All patients with UIAs that are decided to be treated either with endovascular or microsurgical treatments due to several reasons, such as aneurysm size above 4 mm, patient's decision

Exclusion Criteria:

* Prior history of Subarachnoid Hemorrhage (SAH)
* Prior history of intracranial aneurysm
* Severe comorbidities that impact the mental health of the patients, such severe psychiatric disease, and chronic end stage diseases
* Traumatic, mycotic, dissecting, or fusiform aneurysms
* Patients with communication barriers (does not include foreign language), developmental disability, or psychiatric illness that prevent understanding of the questions required to complete assessments
* Patients with any physical disabilities or handicaps

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 6 months
  The number of participants demonstrating anxiety will be determined using the Hospital Anxiety and Depression Scale (HADS) assessment tool. HADS is a widely used tool to evaluate anxiety and depression levels and is composed of 14 items in total, 7 items for anxiety and 7 for depression. The 7 anxiety subscale items are to be answered subjectively by patients using a four-point Likert scale (0-3) with a possible scoring range of 0-21 for anxiety. The number of participants with HADS scores of 8 and above will be considered to demonstrate positive signs of anxiety.

SECONDARY OUTCOMES:
Anxiety | 18 months
  The number of participants demonstrating anxiety will be determined using the Hospital Anxiety and Depression Scale (HADS) assessment tool. HADS is a widely used tool to evaluate anxiety and depression levels and is composed of 14 items in total, 7 items for anxiety and 7 for depression. The 7 anxiety subscale items are to be answered subjectively by patients using a four-point Likert scale (0-3) with a possible scoring range of 0-21 for anxiety. The number of participants with HADS scores of 8 and above will be considered to demonstrate positive signs of anxiety.
Depression | 6 months and 18 months
  The number of participants demonstrating depression will be determined using the Hospital Anxiety and Depression Scale (HADS) assessment tool. HADS is a widely used tool to evaluate anxiety and depression levels and is composed of 14 items in total, 7 items for anxiety and 7 for depression. The 7 depression subscale items are to be answered subjectively by patients using a four-point Likert scale (0-3) with a possible scoring range of 0-21 for depression. The number of participants with HADS scores of 8 and above will be considered to demonstrate positive signs of depression.
Aneurysm rupture | 6 months and 18 months
  The number of participants with any recorded event of aneurysm rupture during the follow-up periods of observed or treated Unruptured Intracranial Aneurysm (UIA) will be determined.
Significant Aneurysm Growth | 6 months and 18 months
  The number of participants demonstrating significant aneurysm growth during the follow-up periods will be determined. Significant aneurysm growth is defined as any aneurysm growth of >= 3 millimeters of observed or treated UIA.
Change in Neurologic Status | 6 months and 18 months
  The number of participants with change in neurologic status will be determined using the National Institute of Health (NIH) Stroke Scale/Score (NIHSS). The NIHSS is a 15-item neurological examination with each item scored on a 3- to 5-point scale, with 0 as normal. Scores range from 0-42 and there is an allowance for untestable items. Progressive increase in NIHSS score by 2 or more points after the procedure and through study completion will be considered as a bad outcome.
Functional Outcome Status | 6 months and 18 months
  The number of participants demonstrating favorable functional outcome status will be assessed using a modified Rankin Scale (mRS) score. Participants with scores ranging from 0 (no disability) to 2 (slight disability) will be considered to have a favorable functional outcome status. Participants with mRS scores ranging from 3 (Moderate disability) to 5 (severe disability) will be considered to have an unfavorable functional outcome status.
Acute adverse events | During admission
  The number of acute adverse events during hospital admission will be tabulated. Acute adverse events will encompass management and procedure-related complications. Increased incidence of procedure-related complications portends more unfavorable outcomes.
Delayed adverse events | 3 months
  The number of delayed adverse events will be tabulated. Delayed adverse events will encompass management and procedure-related complications. Increased incidence of procedure-related complications portends more unfavorable outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: David J Altschul, MD, Principal Investigator — Associate Professor at The Leo M. Davidoff Department of Neurological Surgery at Montefiore
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Player MS, Peterson LE. Anxiety disorders, hypertension, and cardiovascular risk: a review. Int J Psychiatry Med. 2011;41(4):365-77. doi: 10.2190/PM.41.4.f. PMID 22238841
- [Background] Lemos M, Roman-Calderon JP, Calle G, Gomez-Hoyos JF, Jimenez CM. Personality and anxiety are related to health-related quality of life in unruptured intracranial aneurysm patients selected for non-intervention: A cross sectional study. PLoS One. 2020 Mar 12;15(3):e0229795. doi: 10.1371/journal.pone.0229795. eCollection 2020. PMID 32163437
- [Background] Hop JW, Rinkel GJ, Algra A, van Gijn J. Case-fatality rates and functional outcome after subarachnoid hemorrhage: a systematic review. Stroke. 1997 Mar;28(3):660-4. doi: 10.1161/01.str.28.3.660. PMID 9056628
- [Background] Hop JW, Rinkel GJ, Algra A, van Gijn J. Quality of life in patients and partners after aneurysmal subarachnoid hemorrhage. Stroke. 1998 Apr;29(4):798-804. doi: 10.1161/01.str.29.4.798. PMID 9550514
- [Background] Giordan E, Sorenson TJ, Brinjikji W, Vine R, Lanzino G. Risk factors for growth of conservatively managed unruptured intracranial aneurysms. Acta Neurochir (Wien). 2018 Dec;160(12):2419-2423. doi: 10.1007/s00701-018-3729-z. Epub 2018 Nov 11. PMID 30415386
- [Background] van der Schaaf IC, Brilstra EH, Rinkel GJ, Bossuyt PM, van Gijn J. Quality of life, anxiety, and depression in patients with an untreated intracranial aneurysm or arteriovenous malformation. Stroke. 2002 Feb;33(2):440-3. doi: 10.1161/hs0202.102335. PMID 11823649
- [Background] Burckhardt CS, Anderson KL. The Quality of Life Scale (QOLS): reliability, validity, and utilization. Health Qual Life Outcomes. 2003 Oct 23;1:60. doi: 10.1186/1477-7525-1-60. PMID 14613562
- [Background] Stern AF. The hospital anxiety and depression scale. Occup Med (Lond). 2014 Jul;64(5):393-4. doi: 10.1093/occmed/kqu024. No abstract available. PMID 25005549
- [Background] Zhai XD, Yu JX, Ma YJ, Xiang SS, Li GL, He C, Hu P, Zhang HQ. Prevalence of and risk factors for anxiety and depression in Chinese patients with unruptured intracranial aneurysms treated by endovascular intervention. BMC Psychiatry. 2020 Sep 3;20(1):430. doi: 10.1186/s12888-020-02834-3. PMID 32883243
- [Background] Solheim O, Eloqayli H, Muller TB, Unsgaard G. Quality of life after treatment for incidental, unruptured intracranial aneurysms. Acta Neurochir (Wien). 2006 Aug;148(8):821-30; discussion 830. doi: 10.1007/s00701-006-0804-7. Epub 2006 Jun 23. PMID 16791435
- [Background] Preiss M, Netuka D, Koblihova J, Bernardova L, Charvat F, Benes V. Cognitive functions before and 1 year after surgical and endovascular treatment in patients with unruptured intracranial aneurysms. Br J Neurosurg. 2012 Aug;26(4):514-6. doi: 10.3109/02688697.2011.645915. Epub 2012 Jan 19. PMID 22260815
- [Background] Li Y, Dai W, Zhang J. Anxiety, depression and quality of life in patients with a treated or untreated unruptured intracranial aneurysm. J Clin Neurosci. 2017 Nov;45:223-226. doi: 10.1016/j.jocn.2017.07.019. Epub 2017 Aug 1. PMID 28778800
- [Background] Buijs JE, Greebe P, Rinkel GJ. Quality of life, anxiety, and depression in patients with an unruptured intracranial aneurysm with or without aneurysm occlusion. Neurosurgery. 2012 Apr;70(4):868-72. doi: 10.1227/NEU.0b013e3182367295. PMID 21937934
- [Background] Brilstra EH, Rinkel GJ, van der Graaf Y, van Rooij WJ, Algra A. Treatment of intracranial aneurysms by embolization with coils: a systematic review. Stroke. 1999 Feb;30(2):470-6. doi: 10.1161/01.str.30.2.470. PMID 9933290
- [Background] International Study of Unruptured Intracranial Aneurysms Investigators. Unruptured intracranial aneurysms--risk of rupture and risks of surgical intervention. N Engl J Med. 1998 Dec 10;339(24):1725-33. doi: 10.1056/NEJM199812103392401. PMID 9867550
- [Background] Raaymakers TW, Rinkel GJ, Limburg M, Algra A. Mortality and morbidity of surgery for unruptured intracranial aneurysms: a meta-analysis. Stroke. 1998 Aug;29(8):1531-8. doi: 10.1161/01.str.29.8.1531. PMID 9707188
- [Background] Curtis BM, O'Keefe JH Jr. Autonomic tone as a cardiovascular risk factor: the dangers of chronic fight or flight. Mayo Clin Proc. 2002 Jan;77(1):45-54. doi: 10.4065/77.1.45. PMID 11794458
- [Background] Tada Y, Wada K, Shimada K, Makino H, Liang EI, Murakami S, Kudo M, Kitazato KT, Nagahiro S, Hashimoto T. Roles of hypertension in the rupture of intracranial aneurysms. Stroke. 2014 Feb;45(2):579-86. doi: 10.1161/STROKEAHA.113.003072. Epub 2013 Dec 26. PMID 24370755